CLINICAL TRIAL: NCT01482234
Title: TXT Me: Texting Motivational Messages Encouraging Adolescent Physical Activity
Brief Title: Text Messages and Physical Activity Among Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Deborah Thompson, Associate Professor of Pediatrics, Baylor College of Medicine
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: H-27537; R21HD066305 (NIH)
Record Dates: First submitted 2011-11-28; First posted 2011-11-30 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Physical Activity
Keywords: physical activity; exercise; walking; pedometers; goal setting; text messages; motivation; intrinsic motivation; extrinsic motivation; self determination theory; prompts
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- pedometers only (Experimental): Participants randomized to this arm will receive pedometers only. They will participate in baseline and 3 months data collection.
  Interventions: Behavioral: TXT Me
- pedometers + prompts (Experimental): Participants randomized to this arm will receive pedometers plus a weekly prompt to set a step goal. They will participate in baseline and 3 months data collection.
  Interventions: Behavioral: TXT Me
- pedometer + prompt + messages (Experimental): Participants randomized to this arm will receive pedometers, weekly prompts, and 6 motivational text messages a week. They will participate in baseline and 3 months data collection.
  Interventions: Behavioral: TXT Me
- Control (No Intervention): Participants randomized to this group will participate in data collection only; they will not receive an intervention.

INTERVENTIONS:
Behavioral: TXT Me — text messages, physical activity, self determination theory, extrinsic motivation, intrinsic motivation, pedometers, walking, prompts
  Arms: pedometer + prompt + messages; pedometers + prompts; pedometers only

SUMMARY:
The purpose of this study is to assess whether text messages can be used as a way to increase the amount of physical activity teens get each day.

DETAILED DESCRIPTION:
This research will develop an innovative intervention that promotes physical activity to 14-17 year olds (roughly high school aged youth). It is guided by Self Determination Theory and seeks to enhance adolescents' feelings of physical activity autonomy, competence, and relatedness, key psychological needs related to motivation to be physically active. The physical activity to be promoted is walking, which has broad appeal and can be performed as part of usual-day activities. Since youth are heavy users of cell phones and texting, the intervention will send theoretically-grounded text messages designed to enhance physical activity.

ELIGIBILITY:
Inclusion Criteria:

* 14-17 years old
* access to a computer with high speed internet access
* home email address
* cell phone that can send/receive text messages
* text message plan
* fluent in English

Exclusion Criteria:

* mental or physical limitations that impair ability to fully participate in the program and/or complete baseline and post assessment data collection.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2012-02; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
physical activity | 3 months
  physical activity will be assessed for 7 days at each data collection period; accelerometers will be used to assess physical activity amount and intensity

SECONDARY OUTCOMES:
Psychological need satisfaction in exercise | 3 months
  This scale will be used to assess psychological needs related to exercise - autonomy, relatedness, and competence
Behavioral Regulation in Exercise | 3 months
  This scale will be used to assess motivation for exercise
Satisfaction | 3 months
  Satisfaction with the study will be assessed using standard questions

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Thompson, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Derived] Thompson D, Cantu D, Ramirez B, Cullen KW, Baranowski T, Mendoza J, Anderson B, Jago R, Rodgers W, Liu Y. Texting to Increase Adolescent Physical Activity: Feasibility Assessment. Am J Health Behav. 2016 Jul;40(4):472-83. doi: 10.5993/AJHB.40.4.9. PMID 27338994
- [Derived] Thompson D, Cantu D, Bhatt R, Baranowski T, Rodgers W, Jago R, Anderson B, Liu Y, Mendoza JA, Tapia R, Buday R. Texting to Increase Physical Activity Among Teenagers (TXT Me!): Rationale, Design, and Methods Proposal. JMIR Res Protoc. 2014 Mar 12;3(1):e14. doi: 10.2196/resprot.3074. PMID 24622344